CLINICAL TRIAL: NCT02289950
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Assess the Efficacy and Safety of Farletuzumab (MORAb 003) in Combination With Carboplatin Plus Paclitaxel or Carboplatin Plus Pegylated Liposomal Doxorubicin (PLD) in Subjects With Low CA125 Platinum-Sensitive Ovarian Cancer
Brief Title: A Study to Assess the Efficacy and Safety of Farletuzumab (MORAb 003) in Combination With Carboplatin Plus Paclitaxel or Carboplatin Plus Pegylated Liposomal Doxorubicin (PLD) in Participants With Low CA125 Platinum-sensitive Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MORAb-003-011
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Platinum-Sensitive Ovarian Cancer in First Relapse
Keywords: Ovarian Cancer in in first relapse; Platinum-Sensitive
MeSH Terms: interventions — farletuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Farletuzumab (Experimental): All participants will receive a loading dose for the first 2 weeks of 10 milligram per kilogram (mg/kg) farletuzumab, followed by 5 mg/kg weekly farletuzumab administered intravenously (IV).
  Interventions: Drug: Farletuzumab
- Placebo (Placebo Comparator): All subjects will receive placebo weekly, administered intravenously (IV).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Farletuzumab — Farletuzumab will be administered intravenously (IV) weekly
  Arms: Farletuzumab
Drug: Placebo — Placebo will be administered intravenously (IV) weekly
  Arms: Placebo

SUMMARY:
MORAb-003-011 is a global, multicenter, double-blind, randomized placebo-controlled study to assess the safety and efficacy of farletuzumab in combination with standard chemotherapy in subjects with low cancer antigen 125 (CA125) platinum-sensitive ovarian cancer in first relapse.

DETAILED DESCRIPTION:
Participants will be enrolled into 1 of 2 chemotherapy treatment arms at the investigator's discretion: carboplatin plus paclitaxel or carboplatin plus Pegylated Liposomal Doxorubicin (PLD), and then randomized in a 2:1 ratio to receive weekly farletuzumab 5 mg/kg or placebo (ie, Test Article). All participants will receive a loading dose for the first 2 weeks of 10 mg/kg Test Article (farletuzumab or placebo). Participants will be stratified at randomization by individual chemotherapy treatment regimen (targeted 1:1 ratio) and platinum-free interval following first-line therapy (6 to 12 months vs greater than 12 to 36 months).

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects who are at least 18 years of age at the time of informed consent
2. CA125 less than or equal to 3 x upper limit of normal (ULN) [105 units per millilitre (U/mL)] confirmed within 2 weeks of randomization using a centralized laboratory assay
3. A histologically confirmed diagnosis of high-grade serous epithelial ovarian cancer including primary peritoneal and fallopian tube malignancies; all other histologies, including mixed histology, are excluded
4. Have been treated with debulking surgery and a first-line platinum-based chemotherapy regimen
5. Maintenance therapy during the first platinum-free interval is allowed; however, the last dose must have been at least 21 days prior to Randomization.
6. Must be in a first relapse and have evaluable disease by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scan, according to RECIST 1.1 (subjects with measurable disease per RECIST 1.1 or radiographically visible and evaluable disease). Subjects with only ascites or pleural effusion are excluded.
7. Must have relapsed radiographically between 6 months and 36 months of completion of first-line platinum chemotherapy
8. Must be a candidate for treatment with either carboplatin plus paclitaxel or carboplatin plus PLD with no medical contraindications present as outlined in the product labels for the selected regimen to be used in this study
9. Have a life expectancy of at least 6 months, as estimated by the investigator
10. Other significant medical conditions must be well-controlled and stable in the opinion of the investigator for at least 30 days prior to Randomization
11. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
12. Subjects being enrolled to receive paclitaxel plus carboplatin treatment must have neuropathic function (sensory and motor less than or equal to Grade 2 according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v4.03 (2010)
13. Laboratory results within the 2 weeks prior to Randomization must be as follows:

    * Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L
    * Platelet count greater than or equal to 100 x 10^9/L
    * Hemoglobin greater than or equal to 9 g/dL
    * Creatinine less than 1.5 x ULN (CTCAE Grade 1)
    * Bilirubin less than 1.5 x ULN (CTCAE Grade 1)
    * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) less than 3 x ULN
    * Alkaline Phosphatase less than 2.5 x ULN (CTCAE Grade 1)
    * Baseline albumin greater than or equal to Lower Limit of Normal
14. Subjects of childbearing potential must be surgically sterile or consent to use a medically acceptable method of contraception throughout the study period. All females will be considered to be of childbearing potential unless they are postmenopausal (eg, amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing). If a patient of childbearing potential is neither surgically sterile nor postmenopausal, a highly-effective contraceptive method (ie, a method that can achieve a failure rate of less than 1 percent (%) per year when used consistently and correctly) must start either before or at Screening and continue throughout the entire study period and for 6 months after the last dose of Test Article is administered. Pregnant and/or lactating females are excluded

Exclusion Criteria:

1. Known central nervous system (CNS) tumor involvement
2. Evidence of other active invasive malignancy requiring treatment other than surgery in the past 3 years
3. Clinically significant heart disease (eg, congestive heart failure of New York Heart Association Class 3 or 4 angina, not well controlled by medication, or myocardial infarction within 6 months)
4. Electrocardiogram (ECG) demonstrating clinically significant arrhythmias that are not adequately medically managed (Note: subjects with chronic atrial arrhythmia, ie, atrial fibrillation or paroxysmal supraventricular tachycardia [SVT], are eligible)
5. Active serious systemic disease, including active bacterial or fungal infection
6. Active viral hepatitis or active human immunodeficiency virus (HIV) infection. Asymptomatic positive serology is not exclusionary.
7. Other concurrent immunotherapy (eg, immunosuppressants or chronic use of systemic corticosteroids, with the exception that low-dose corticosteroids [50 mg/day prednisone or equivalent corticosteroid] are allowed; these should be discussed with the Medical Monitor)
8. Known allergic reaction to a prior monoclonal antibody therapy or have any documented Anti-Drug Antibody (ADA) response; additionally known allergic reaction to the concomitant chemotherapies selected by the investigator for planned treatment in this study unless desensitization is planned
9. Previous treatment with farletuzumab or other folate receptor targeting agents
10. Previous treatment with cancer vaccine therapy
11. For subjects being enrolled to receive PLD plus carboplatin, prior treatment with anthracyclines or anthracenodiones
12. Breast-feeding, pregnant, or likely to become pregnant during the study
13. Any medical or other condition that, in the opinion of the investigator, would preclude the subject's participation in a clinical study including medical contraindications as outlined in the product labels for the chemotherapies selected by the investigator for planned treatment in this study
14. Patients who have had secondary debulking surgery or any second line therapy
15. Currently enrolled in another clinical study or used any investigational drug or device within 30 days (or 5 x half-life for investigational drugs where the half-life is known) preceding informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (35):
  - Phoenix, Arizona
  - Los Angeles, California
  - Orange, California
  - Roseville, California
  - Sacramento, California
  - Aurora, Colorado
  - Miami, Florida
  - Miramar, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Grand Island, Nebraska
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Austin, Texas
  - Annandale, Virginia
  - Charlottesville, Virginia
- Belgium (6):
  - Edegem, Antwerpen
  - Brussels, Brussels Capital
  - Hasselt, Limburg
  - Ghent, Oost-Vlaanderen
  - Leuven
  - Liège
- Germany (5):
  - Ulm, Baden-Wurttemberg
  - Chemnitz, Saxony
  - Berlin
  - Dresden
  - Essen
- Italy (8):
  - Bari, Apulia
  - Napoli, Campania
  - Rome, Lazio
  - Avellino
  - Bologna
  - Milan
  - Napoli
  - Perugia
- Japan (8):
  - Chūōku
  - Hidaka
  - Kashiwa
  - Kōtoku
  - Kurume
  - Matsuyama
  - Minatoku
  - SuntoGun
- Spain (4):
  - Palma de Mallorca, Balearic Islands
  - Córdoba, Córdoba
  - Madrid
  - Sabadell
- United Kingdom (2):
  - Plymouth, Devon
  - London

REFERENCES:
- [Derived] Herzog TJ, Pignata S, Ghamande SA, Rubio MJ, Fujiwara K, Vulsteke C, Armstrong DK, Sehouli J, Coleman RL, Gabra H, Scambia G, Monk BJ, Arranz JA, Ushijima K, Hanna R, Zamagni C, Wenham RM, Gonzalez-Martin A, Slomovitz B, Jia Y, Ramsay L, Tewari KS, Weil SC, Vergote IB. Randomized phase II trial of farletuzumab plus chemotherapy versus placebo plus chemotherapy in low CA-125 platinum-sensitive ovarian cancer. Gynecol Oncol. 2023 Mar;170:300-308. doi: 10.1016/j.ygyno.2023.01.003. Epub 2023 Feb 7. PMID 36758420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 60 investigative sites in the United states, Belgium, Germany, Italy, Spain, United Kingdom and Japan from 19 March 2015 to 13 August 2020.
Pre-assignment Details: A total of 332 participants were screened, of which 118 were screen failures and 214 were randomized out of which 211 were treated. .
Groups:
- Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD: Participants received either carboplatin (area under the concentration-time curve [AUC] 5) plus paclitaxel 175 milligrams per square meter (mg/m^2) intravenously (IV) every 3 weeks or carboplatin (AUC 5) plus pegylated liposomal doxorubicin (PLD) 30 mg/m^2 IV every 4 weeks in combination with farletuzumab loading dose of 10 milligram per kilogram (mg/kg) for the first 2 weeks, followed by 5 mg/kg every week thereafter administered up to maximum of 8 cycles at the investigator's discretion. Participants who completed combination treatment phase and participants who experienced intolerable toxicity to chemotherapy in combination treatment phase continued to receive maintenance treatment with farletuzumab 5 mg/kg every week alone up to maximum of 64 cycles or until disease progression was confirmed by radiographic assessment, or participant discontinued treatment for any other reason.
- Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD: Participants received either carboplatin (AUC 5) plus paclitaxel 175 mg/ m^2 IV every 3 weeks or carboplatin (AUC 5) plus PLD 30 mg/ m^2 IV every 4 weeks in combination with placebo loading dose of 10 mg/kg for the first 2 weeks, followed by 5 mg/kg every week thereafter administered up to maximum of 8 cycles at the investigator's discretion. Participants who completed combination treatment phase and participants who experienced intolerable toxicity to chemotherapy in combination treatment phase continued to receive maintenance treatment with placebo 5 mg/kg every week alone up to maximum of 64 cycles or until disease progression was confirmed by radiographic assessment, or subject discontinued treatment for any other reason.
Period: Overall Study
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD
Started (214) | 142 | 72
Treated | 140 (1 participant randomized to placebo group but was treated with farletuzumab, and was analyzed in the farletuzumab group in safety analysis set.) | 71
Completed | 0 | 0
Not Completed | 142 | 72
Not completed — Progressive disease by RECIST 1.1 | 99 | 52
Not completed — Progressive disease by Clinical Assessment | 4 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 9 | 3
Not completed — Subject chose to discontinue therapy but will continue to survival follow-up | 9 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Test article held for greater than 28 days | 0 | 1
Not completed — Adverse Event | 11 | 3
Not completed — Death | 1 | 1
Not completed — Other | 5 | 2
Not completed — Not Treated | 2 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) Population (the Full Analysis Set) included all randomized participants according to the assigned treatment by interactive response technology (IRT) system.
Groups:
- Total: Total of all reporting groups
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD | Total
Number analyzed (Participants) | 142 | 72 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (10.74) | 62.9 (10.50) | 62.3 (10.64)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females | 141 | 72 | 213
  Unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 3 | 15
  Not Hispanic or Latino | 126 | 68 | 194
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 8 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 117 | 62 | 179
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time (in months) from the date of randomization of a participant to the date of first observation of progression or date of death, whatever the cause. PFS was assessed based on the investigators' assessments utilizing Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Disease progression (PD) was defined as at least a 20 percent (%) increase or 5 millimeter (mm) increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. PFS was estimated and analyzed using Kaplan-Meier method.
Time Frame: From the date of randomization to the date of first documentation of PD, or date of death, whichever occurs first up to approximately 5 years 5 months
Population: The ITT Population (Full Analysis Set) included all randomized participants according to the assigned treatment by IRT system.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD
Number analyzed (Participants) | 142 | 72
Months | 11.73 [10.22 to 13.60] | 10.78 [9.49 to 13.17]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death. Participants were censored at the date of last known to be alive. OS was analyzed using Kaplan-Meier method.
Time Frame: From the date of randomization until the date of death (up to approximately 5 years 5 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD
Number analyzed (Participants) | 142 | 72
Months | 43.07 [37.13 to NA] — Here, NA means that the upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of events. | 42.45 [37.85 to NA] — Here, NA means that the upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of events.

3. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: BOR was defined as the best response of complete response (CR) or partial response (PR) or stable disease (SD) for greater than or equal to(>=)6 months recorded from the start of the treatment until PD or death, whichever occurred first based on investigator assessment per RECIST v1.1. CR:disappearance of all target and non-target lesions. All pathological (whether target or non-target) must have a reduction in their short axis less than(<)10 mm. PR:at least a 30% decrease in the sum of diameter (SOD) of target lesions, taking as reference the baseline sum diameters. SD:neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD. PD was defined as at least 20% increase (including an absolute increase of at least 5mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From first dose of study drug (Baseline) up to approximately 5 years 5 months
Population: Tumor Response Evaluable Analysis Set included all randomized participants who received at least 1 dose of study drug and who had a baseline and at least 1 on treatment tumor assessment performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD
Number analyzed (Participants) | 138 | 68
Participants
  Complete Response | 24 | 15
  Partial Response | 72 | 35
  Stable Disease | 36 | 17

4. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR was defined as the time (in months) from the date of randomization to the date of first observation of response (PR or CR) (whichever status was recorded first). TTR was assessed based on investigator assessment utilizing RECIST 1.1. CR: disappearance of all target and non-target lesions. All pathological (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD.
Time Frame: From the date of randomization until date of first observation of response (CR or PR) up to approximately 5 years 5 months
Population: Tumor Response Evaluable Analysis Set included all randomized participants who received at least 1 dose of study drug and who had a baseline and at least 1 on treatment tumor assessment performed. Here "overall number of participants analyzed" signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD
Number analyzed (Participants) | 96 | 50
months | 2.69 [1.74 to 2.83] | 2.53 [1.48 to 2.69]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time (in months) from the date of first observation of response (PR or CR) to the date of the first observation of progression based on the investigator's assessment utilizing RECIST 1.1, or date of death, whatever the cause. CR: disappearance of all target and non-target lesions. All pathological (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30 % decrease in the SOD of target lesions, taking as reference the baseline sum diameters. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From date of the first observation of CR or PR until the date of first observation of progression or date of death up to approximately 5 years 5 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD
Number analyzed (Participants) | 96 | 50
months | 10.12 [8.54 to 11.47] | 8.51 [6.31 to 10.97]

6. Secondary Outcome: Percentage of Participants Achieving Each Second Platinum-Free Interval Stratified by First Platinum-Free Interval
Description: Percentage of participants achieving each second platinum-free interval (<6 months, 6-12 months, greater than [>] 12-36 months, and >36 months) stratified by first platinum-free interval (6 to 12 months and >12 to 36 months) was reported. First platinum-free interval was defined as the date of completion of previous platinum-based chemotherapy until the date of first relapse (that is, first observation of progression). The date of first relapse was the progression date. Second platinum-free interval was defined as the date of completion of platinum-based chemotherapy (last dosing date) during the study until the date of progression or death (or censoring, if applicable).
Time Frame: From the date of randomization to the date of first relapse (or first observation of progression/death) up to approximately 5 year 5 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD
Number analyzed (Participants) | 142 | 72
percentage of participants
  Second platinum free interval (<6 months): First platinum free interval (6 to 12 months) | 71.2 [57.92 to 82.24] | 63.3 [43.86 to 80.07]
  Second platinum free interval (6-12 months): First platinum free interval (6 to 12 months) | 6.8 [1.88 to 16.46] | 23.3 [9.93 to 42.28]
  Second platinum free interval (>12-36 months): First platinum free interval (6 to 12 months) | 16.9 [8.44 to 28.97] | 10.0 [2.11 to 26.53]
  Second platinum free interval (>36 months): First platinum free interval (6 to 12 months) | 0.00 [0.00 to 6.06] | 0.0 [0.00 to 11.57]
  Second platinum free interval (<6 months): First platinum free interval (>12 to 36 months) | 42.2 [31.40 to 53.51] | 52.4 [36.42 to 68.00]
  Second platinum free interval (6-12 months): First platinum free interval (>12 to 36 months) | 33.7 [23.72 to 44.95] | 28.6 [15.72 to 44.58]
  Second platinum free interval (>12-36 months): First platinum free interval (>12 to 36 months) | 20.5 [12.41 to 30.76] | 16.7 [6.97 to 31.36]
  Second platinum free interval (>36 months): First platinum free interval (>12 to 36 months) | 0.0 [0.00 to 4.35] | 0.0 [0.00 to 8.41]

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study treatment (up to approximately 5 years 5 months)
Description: Deaths that happened anytime during the study (including those during the treatment and after treatment discontinuation) are reported in this section.
Arm/Group | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD
All-Cause Mortality (participants affected / at risk) | 1/141 | 2/70
Serious Adverse Events (participants affected / at risk) | 42/141 | 18/70
Other Adverse Events (participants affected / at risk) | 140/141 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD (N=141) | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD (N=70)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (9) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 5 (6) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (13) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (2) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Farletuzumab 5 mg/kg + Carboplatin/Paclitaxel or Carboplatin/PLD (N=141) | Placebo + Carboplatin/Paclitaxel or Carboplatin/PLD (N=70)
Anaemia (Blood and lymphatic system disorders) | 76 (208) | 36 (121)
Neutropenia (Blood and lymphatic system disorders) | 55 (225) | 24 (82)
Leukopenia (Blood and lymphatic system disorders) | 21 (74) | 7 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 42 (109) | 19 (86)
Abdominal discomfort (Gastrointestinal disorders) | 9 (14) | 9 (11)
Abdominal distension (Gastrointestinal disorders) | 9 (12) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 39 (65) | 22 (34)
Abdominal pain upper (Gastrointestinal disorders) | 17 (19) | 12 (17)
Constipation (Gastrointestinal disorders) | 58 (93) | 31 (53)
Diarrhoea (Gastrointestinal disorders) | 48 (83) | 27 (63)
Dry mouth (Gastrointestinal disorders) | 9 (9) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 12 (15) | 10 (14)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (18) | 5 (6)
Nausea (Gastrointestinal disorders) | 95 (187) | 45 (110)
Stomatitis (Gastrointestinal disorders) | 44 (66) | 24 (51)
Vomiting (Gastrointestinal disorders) | 43 (74) | 27 (56)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 8 (8) | 6 (9)
Vision blurred (Eye disorders) | 7 (7) | 5 (5)
Asthenia (General disorders) | 33 (90) | 14 (42)
Chills (General disorders) | 6 (9) | 5 (5)
Fatigue (General disorders) | 69 (112) | 35 (55)
Influenza like illness (General disorders) | 8 (10) | 4 (5)
Malaise (General disorders) | 9 (14) | 9 (11)
Oedema peripheral (General disorders) | 16 (21) | 12 (19)
Peripheral swelling (General disorders) | 4 (4) | 4 (4)
Pyrexia (General disorders) | 23 (37) | 11 (16)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 5 (6)
Cystitis (Infections and infestations) | 6 (9) | 4 (5)
Influenza (Infections and infestations) | 9 (12) | 7 (9)
Nasopharyngitis (Infections and infestations) | 22 (34) | 14 (26)
Sinusitis (Infections and infestations) | 10 (11) | 8 (11)
Upper respiratory tract infection (Infections and infestations) | 23 (29) | 6 (8)
Urinary tract infection (Infections and infestations) | 18 (24) | 16 (32)
Alanine aminotransferase increased (Investigations) | 7 (10) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 10 (16) | 4 (4)
Neutrophil count decreased (Investigations) | 44 (165) | 18 (90)
Platelet count decreased (Investigations) | 27 (83) | 11 (46)
White blood cell count decreased (Investigations) | 34 (127) | 14 (68)
Decreased appetite (Metabolism and nutrition disorders) | 28 (43) | 18 (32)
Dehydration (Metabolism and nutrition disorders) | 13 (21) | 7 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (18) | 6 (6)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 (12) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (49) | 4 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 (33) | 7 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 (52) | 15 (27)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (24) | 18 (24)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 4 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (9) | 11 (17)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (15) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (19) | 7 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (22) | 12 (18)
Dizziness (Nervous system disorders) | 22 (40) | 13 (19)
Dysgeusia (Nervous system disorders) | 15 (22) | 12 (17)
Headache (Nervous system disorders) | 49 (77) | 27 (61)
Paraesthesia (Nervous system disorders) | 11 (14) | 8 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (31) | 14 (21)
Anxiety (Psychiatric disorders) | 15 (18) | 5 (5)
Depression (Psychiatric disorders) | 6 (6) | 6 (16)
Insomnia (Psychiatric disorders) | 15 (17) | 8 (11)
Dysuria (Renal and urinary disorders) | 11 (16) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 43 (65) | 16 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (47) | 9 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 7 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (29) | 15 (19)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5) | 9 (10)
Erythema (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (4)
Nail discolouration (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 (13) | 9 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (17) | 9 (14)
Rash (Skin and subcutaneous tissue disorders) | 24 (38) | 13 (15)
Hot flush (Vascular disorders) | 4 (4) | 9 (17)
Hypertension (Vascular disorders) | 7 (10) | 5 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT02289950/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT02289950/SAP_001.pdf